CLINICAL TRIAL: NCT07213856
Title: Nutritional Intervention for Constipation Symptoms in Patients With Parkinson's Disease: A Randomized Clinical Trial
Brief Title: Nutritional Intervention for Constipation Symptoms in Patients With Parkinson's Disease
Acronym: NUTRI-GUT-PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0374
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Parkinsons Disease (PD); Constipation - Functional
Keywords: Microbiota; Diet; Diet, Protein-Restricted; Diet Therapy; Diet, Healthy; Nutrition Therapy; Constipation; Non-Motor Symptoms; Nutritionists
MeSH Terms: conditions — Parkinson Disease; Constipation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Intervention Group (Experimental): Participants will receive a tailored diet plan made by a registered dietitian, with follow-ups for 3 months. The plan is based on Dietary Reference Intakes and adapted to Parkinson's disease and constipation management guidelines.
  Interventions: Behavioral: Dietitian-Guided Nutritional Intervention
- Control Group (No Intervention): Participants will not receive individualized nutritional support during the study period. They will receive the dietary guidance only after the end of the study (3 months).

INTERVENTIONS:
Behavioral: Dietitian-Guided Nutritional Intervention — Participants receive a diet plan and nutritional counseling provided by a registered dietitian, based on a standardized protocol aligned with the Dietary Reference Intakes (DRIs) and adapted for the management of Parkinson's disease and constipation. The intervention includes follow-ups with the dietitian over a 3-month period.
  Other Names: Diet plan
  Arms: Nutritional Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate whether a dietitian-guided nutritional intervention can improve constipation symptoms in people with Parkinson's disease (PD). The main questions it aims to answer are:

* Can a dietitian-guided nutritional intervention increase the number of weekly bowel movements in individuals with PD and functional constipation?
* Can this intervention positively influence gut microbiota composition, dietary intake, and nutritional status?

Researchers will compare the intervention group to a control group that will receive general dietary guidance only after the study period, to see if the intervention leads to improvements in bowel function and related health outcomes.

Participants will:

* Follow a diet plan developed by a dietitian, based on dietary reference intakes and tailored to the needs of individuals with PD and constipation
* Participate in follow-up sessions with the dietitian for 3 months
* Complete assessments at baseline, midpoint, and end of the intervention to evaluate bowel function, constipation symptoms, gut microbiota, nutritional status, and diet quality

ELIGIBILITY:
Inclusion Criteria:

* Adults with a previous diagnosis of Parkinson's disease
* On a stable dose of levodopa for at least 3 months
* Diagnosis of Functional Constipation by the Rome IV protocol

Exclusion Criteria:

* Diagnosis of atypical or secondary parkinsonism
* Hoehn and Yahr stage greater than 2
* Presence of severe neurological or psychiatric disorders that impair the ability to participate in study procedures
* Previous diagnosis of dementia
* Presence of comorbidities such as active cancer, chronic obstructive pulmonary disease (COPD), heart failure, and/or chronic kidney disease
* History of gastrointestinal cancers, inflammatory bowel diseases, or surgeries involving the gastrointestinal tract
* Constipation secondary to clinical conditions such as hypothyroidism or diabetes mellitus
* Use of opioids
* Use of probiotics or antibiotics in the past 8 weeks
* Continuous use of laxatives in the past 8 weeks
* Presence of severe dysphagia according to the Functional Oral Intake Scale (FOIS)
* Individuals receiving enteral or parenteral nutrition
* Individuals under nutritional follow-up in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in weekly bowel movement frequency | Baseline and 90 days
  Mean change in the number of spontaneous bowel movements per week from baseline to 12 weeks, based on participant-reported bowel diaries.

SECONDARY OUTCOMES:
Change in relative abundance of gut microbial taxa | Baseline and 90 days
  Change in the relative abundance of selected bacterial genera associated with constipation and Parkinson's disease, measured by 16S rRNA sequencing of stool samples.

OTHER OUTCOMES:
Change in dietary intake | Baseline, 45 days and 90 days
  Variation in intake of macronutrients and fiber, assessed through 24h food records.

CONTACTS AND LOCATIONS:
Overall Officials: Maira Rozenfeld Olchik, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Food and Nutrition Board; Committee on the Dietary Reference Intakes for Energy. Dietary Reference Intakes for Energy. Washington (DC): National Academies Press (US); 2023 Jan 17. Available from http://www.ncbi.nlm.nih.gov/books/NBK588659/ PMID 36693139
- [Background] Barichella M, Cereda E, Cassani E, Pinelli G, Iorio L, Ferri V, Privitera G, Pasqua M, Valentino A, Monajemi F, Caronni S, Lignola C, Pusani C, Bolliri C, Faierman SA, Lubisco A, Frazzitta G, Petroni ML, Pezzoli G. Dietary habits and neurological features of Parkinson's disease patients: Implications for practice. Clin Nutr. 2017 Aug;36(4):1054-1061. doi: 10.1016/j.clnu.2016.06.020. Epub 2016 Jul 5. PMID 27406858
- [Background] Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology. 2016 May;150(6):1257-61. doi: 10.1053/j.gastro.2016.03.035. No abstract available. PMID 27147121
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316